CLINICAL TRIAL: NCT01119703
Title: A Phase I, Open-Label Observational Study to Develop a Prospective Predictor of Vaccine Hyporesponse in Healthy Elderly Subjects
Brief Title: Vaccine Hyporesponse in Healthy Elderly Participants (MK-0000-131 AM2)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-131; MK-0000-131 (Other: Merck)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Vaccine Response Impaired
Keywords: Vaccine Hyporesponse
MeSH Terms: interventions — Tetanus Toxoid; Hepatitis B Vaccines; Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cryopreserved peripheral blood mononuclear cells (PBMCs) obtained from whole blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1: Healthy, elderly participants: Healthy participants 65 years old and older.
  Interventions: Biological: Tetanus & Diphtheria booster vaccine (Td); Biological: TwinrixTM [Hepatitis A Inactivated & Hepatitis B (Recombinant) Vaccine]; Biological: Dukoral® Traveler's Diarrhea Vaccine (WC/rBS)
- Arm 2: Healthy, young, participants: Healthy participants 25 to 40 years old.
  Interventions: Biological: Tetanus & Diphtheria booster vaccine (Td); Biological: TwinrixTM [Hepatitis A Inactivated & Hepatitis B (Recombinant) Vaccine]; Biological: Dukoral® Traveler's Diarrhea Vaccine (WC/rBS)

INTERVENTIONS:
Biological: Tetanus & Diphtheria booster vaccine (Td) — Tetanus & Diphtheria booster vaccine (Td), single intramuscular dose
Biological: TwinrixTM [Hepatitis A Inactivated & Hepatitis B (Recombinant) Vaccine] — TwinrixTM [Hepatitis A Inactivated & Hepatitis B (Recombinant) Vaccine], intramuscular, two doses of standard three dose regimen (opposite arms)
Biological: Dukoral® Traveler's Diarrhea Vaccine (WC/rBS) — Dukoral® Traveler's Diarrhea Vaccine, recombinant Cholera toxin B subunit (WC/rBS), standard two oral doses per treatment regimen

SUMMARY:
This study evaluated whether it is possible in healthy elderly participants to generate baseline biomarker-based prediction rules (PdR) for vaccine response (post baseline absolute serum antibody titer) using each of the protocol selected vaccines separately; and examined the rank correlation coefficients of pairs of post vaccination antibody titers within the same elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 25 to 40 years old or 65 years of age or older at the prestudy (screening) visit
* Has no fever on day of screening
* Lacks Hepatitis B surface antigen seroreactivity
* If female 25 to 40 years of age, is not pregnant nor breastfeeding, and agrees to use effective contraception

Exclusion Criteria:

* Has a prior history of Hepatitis B Virus infection
* Has BMI (Body Mass Index) >35
* If female 25 to 40 years of age, is pregnant, or expecting to conceive, donate eggs or breastfeed
* Has received immune globulin and/or blood products within 3 months prior to first dose received
* Has a history of immunosuppression resulting from disease (e.g., malignancy; human immunodeficiency virus [HIV] infection), or is currently taking corticosteroids or other immunosuppressive/cytotoxic therapy (cancer chemotherapy or organ transplantation)
* Has an active neoplastic disease
* Has had any infection including upper respiratory viral syndrome in the 6 weeks prior to planned collection of baseline laboratory samples
* Has received a live virus vaccine or an inactivated vaccine or is scheduled to receive a live virus vaccine or an inactivated vaccine in the period from 6 weeks prior to receipt of the first vaccine through the completion of all study visits

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 25 to 40 years old or 65 years and older
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois St-Maurice, MD, Principal Investigator — Anapharm; Denis Audet, MD, Principal Investigator — Anapharm

RESULTS

PARTICIPANT FLOW:
Groups:
- Younger Participants: Participants 25 to 40 years of age.
- Elderly Participants: Participants 65 years old and older.
Period: Overall Study
Arm/Group | Younger Participants | Elderly Participants
Started | 30 | 144
Completed | 30 | 143
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Younger Participants: Aged 25 to 40 years old
- Elderly Participants: Aged 65 years and older
- Total: Total of all reporting groups
Arm/Group | Younger Participants | Elderly Participants | Total
Number analyzed (Participants) | 30 | 144 | 174
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.9 (3.6) | 70.2 (4.1) | 63.9 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 77 | 95
  Male | 12 | 67 | 79

OUTCOME MEASURES:

1. Primary Outcome: Antibody Titer Responses to Hepatitis B Virus Surface Antigen (HBV sAg) Vaccine, Measured and Predicted Based on Pre-vaccination Biomarkers in Healthy, Elderly Participants.
Description: Healthy elderly participants were simultaneously vaccinated at baseline with hepatitis vaccine, tetanus-diphtheria booster vaccine, and cholera vaccine. Antibody titers to HBV sAg were then measured 1 month after final vaccination, based on enzyme linked immunosorbent assay (ELISA), and are defined as standardized "international units" of reactivity converted from optical densities, transformed to natural log (ln). In order to predict antibody responses blood samples were collected prior to vaccination at baseline, to measure a wide variety of biomarkers by messenger RNA (mRNA) profiling, biochemical and flow cytometric assays. These biomarkers were then used in a machine-learning (random-forest based) model to predict antibody titers, transformed to natural log (ln).
Time Frame: Baseline and 1 month after final vaccination
Population: Healthy participants 65 years of age and older who were treated with all three vaccines, and had their post-vaccination titers measured. Results from comparing titers and biomarker responses between younger and older cohorts are exploratory, and therefore not reported.
Measure: Mean (Standard Deviation); unit: ln International Units
Groups:
- Elderly Participants: Healthy participants 65 years of age and older.
Arm/Group | Elderly Participants
Number analyzed (Participants) | 143
ln International Units
  Predicted Titer | 2.27 (1.24)
  Measured Titer | 2.12 (1.91)
Statistical Analysis 1: Comparison: Elderly Participants; Null hypothesis for Predicted versus Measured Titers states that Coefficient of Determination % (CD%) <= 20%; whereas the alternative hypothesis is > 20%. CD% was obtained by fitting a random forest model to the measured titers, which included all baseline biomarkers as predictors; Test type: Superiority or Other; Coefficient of Determination % = -9.1, 95% CI 2-sided [-13.8 to -0.7] — Crossvalidated; negative values mean that the fitted model performs worse than chance on the test set

2. Primary Outcome: Antibody Titer Responses to Tetanus Booster Vaccine, Measured and Predicted Based on Pre-vaccination Biomarkers in Healthy, Elderly Participants.
Description: Healthy elderly participants were simultaneously vaccinated at baseline with hepatitis vaccine, tetanus-diphtheria booster vaccine, and cholera vaccine. Antibody titers to tetanus were then measured 1 month after final vaccination, based on ELISA, and are defined as standardized "international units" of reactivity converted from optical densities, transformed to natural log (ln). In order to predict antibody responses blood samples were collected prior to vaccination at baseline, to measure a wide variety of biomarkers by mRNA profiling, biochemical and flow cytometric assays. These biomarkers were then used in a machine-learning (random-forest based) model to predict antibody titers, transformed to natural log (ln).
Time Frame: Baseline and 1 month after final vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln International Units
Arm/Group | Elderly Participants
Number analyzed (Participants) | 143
ln International Units
  Predicted Titer | 1.40 (1.24)
  Measured Titer | 1.32 (1.84)
Statistical Analysis 1: Comparison: Elderly Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Coefficient of Determination % = 17.6, 95% CI 2-sided [10.6 to 20.9] — Crossvalidated; negative values mean that the fitted model performs worse than chance on the test set

3. Primary Outcome: Antibody Titer Responses to Reduced Diphtheria Toxin Vaccine, Measured and Predicted Based on Pre-vaccination Biomarkers in Healthy, Elderly Participants.
Description: Healthy elderly participants were simultaneously vaccinated at baseline with hepatitis vaccine, tetanus-diphtheria booster vaccine, and cholera vaccine. Antibody titers to diphtheria were then measured 1 month after final vaccination, based on ELISA, and are defined as standardized "international units" of reactivity converted from optical densities, transformed to natural log (ln). In order to predict antibody responses blood samples were collected prior to vaccination at baseline, to measure a wide variety of biomarkers by mRNA profiling, biochemical and flow cytometric assays. These biomarkers were then used in a machine-learning (random-forest based) model to predict antibody titers, transformed to natural log (ln).
Time Frame: Baseline and 1 month after final vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln International Units
Arm/Group | Elderly Participants
Number analyzed (Participants) | 143
ln International Units
  Predicted Titer | -0.43 (1.25)
  Measured Titer | -0.46 (1.77)
Statistical Analysis 1: Comparison: Elderly Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Coefficient of Determination % = 27.8, 95% CI 2-sided [19.6 to 32.4] — Crossvalidated; negative values mean that the fitted model performs worse than chance on the test set

4. Primary Outcome: Antibody Titer Responses to Oral Cholera Vaccine (WC/rBS), Measured and Predicted Based on Pre-vaccination Biomarkers in Healthy, Elderly Participants.
Description: Healthy elderly participants were simultaneously vaccinated at baseline with hepatitis vaccine, tetanus-diphtheria booster vaccine, and cholera vaccine. Antibody titers to cholera were then measured 3 weeks after final vaccination, based on ELISA, and are defined as standardized "international units" of reactivity converted from optical densities, transformed to natural log (ln). In order to predict antibody responses blood samples were collected prior to vaccination at baseline, to measure a wide variety of biomarkers by mRNA profiling, biochemical and flow cytometric assays. These biomarkers were then used in a machine-learning (random-forest based) model to predict antibody titers, transformed to natural log (ln).
Time Frame: Baseline and 3 weeks after final vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln International Units
Arm/Group | Elderly Participants
Number analyzed (Participants) | 143
ln International Units
  Predicted Titer | 5.24 (0.99)
  Measured Titer | 5.20 (1.55)
Statistical Analysis 1: Comparison: Elderly Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Coefficient of Determination % = 3.3, 95% CI [-2.8 to 8.5] — Crossvalidated; negative values mean that the fitted model performs worse than chance on the test set

5. Primary Outcome: Post-vaccination Antibody Titer Responses to Different Vaccines in Healthy, Elderly, Participants.
Description: Healthy elderly participants were simultaneously vaccinated at baseline with hepatitis vaccine, tetanus-diphtheria booster vaccine, and cholera vaccine. Antibody titers to each of these four antigens were then measured 1 month after each final vaccination (3 weeks for cholera toxin), based on ELISA, and are defined as standardized "international units" of reactivity converted from optical densities, transformed to natural log (ln).
Time Frame: 3 weeks or 1 month after each final vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln International Units
Arm/Group | Elderly Participants
Number analyzed (Participants) | 143
ln International Units
  Hepatitis B | 2.12 (1.91)
  Tetanus | 1.32 (1.84)
  Diphtheria | -0.46 (1.77)
  Cholera | 5.20 (1.55)
Statistical Analysis 1: Comparison: Elderly Participants; Diphtheria versus Hepatitis B; Test type: Superiority or Other; p = 0.66, Fisher's Z-transformation; Spearman's Correlation Coefficient = -0.04, 95% CI 2-sided [-0.2 to 0.13] — Within-participant rank correlation
Statistical Analysis 2: Comparison: Elderly Participants; Diphtheria versus Cholera; Test type: Superiority or Other; p = 0.26, Fisher's Z-transformation; Spearman's Correlation Coefficient = 0.10, 95% CI 2-sided [-0.07 to 0.25] — Within-participant rank correlation
Statistical Analysis 3: Comparison: Elderly Participants; Diphtheria versus Tetanus; Test type: Superiority or Other; p < 0.001, Fisher's Z-transformation; Spearman's Correlation Coefficient = 0.40, 95% CI 2-sided [0.26 to 0.53] — Within-participant rank correlation
Statistical Analysis 4: Comparison: Elderly Participants; Hepatitis B versus Cholera; Test type: Superiority or Other; p = 0.04, Fisher's Z-transformation; Spearman's Correlation Coefficient = -0.17, 95% CI 2-sided [-0.32 to -0.01] — Within-participant rank correlation
Statistical Analysis 5: Comparison: Elderly Participants; Hepatitis B versus Tetanus; Test type: Superiority or Other; p = 0.30, Fisher's Z-transformation; Spearman's Correlation Coefficient = -0.09, 95% CI 2-sided [-0.25 to 0.08] — Within-participant rank correlation
Statistical Analysis 6: Comparison: Elderly Participants; Cholera versus Tetanus; Test type: Superiority or Other; p = 0.36, Fisher's Z-transformation; Spearman's Correlation Coefficient = 0.08, 95% CI 2-sided [-0.09 to 0.24] — Within-participant rank correlation

6. Secondary Outcome: Antibody Titer Responses to Hepatitis B Virus Surface Antigen (HBV sAg) Vaccine, Measured and Predicted Based on Early Post-vaccination Biomarkers in Healthy, Elderly Participants.
Description: Healthy elderly participants were simultaneously vaccinated at baseline with hepatitis vaccine, tetanus-diphtheria booster vaccine, and cholera vaccine. Antibody titers to HBV sAg were then measured 1 month after final vaccination, based on ELISA, and are defined as standardized "international units" of reactivity converted from optical densities, transformed to natural log (ln). In order to predict antibody responses blood samples were collected at 7 days post-baseline vaccination to measure a wide variety of biomarkers by mRNA profiling, biochemical and flow cytometric assays. These biomarkers were then used in a machine-learning (random-forest based) model to predict antibody titers, transformed to natural log (ln).
Time Frame: Day 7 and 1 month after final vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln International Units
Arm/Group | Elderly Participants
Number analyzed (Participants) | 143
ln International Units
  Predicted Titer | 2.25 (1.24)
  Measured Titer | 2.12 (1.91)
Statistical Analysis 1: Comparison: Elderly Participants; Null hypothesis for Predicted versus Measured Titers states that Coefficient of Determination % (CD%) <= 20%; whereas the alternative hypothesis is > 20%. CD% was obtained by fitting a random forest model to the measured titers, which included all Day 7 biomarkers as predictors; Test type: Superiority or Other; Coefficient of Determination % = -9.5, 95% CI 2-sided [-16.6 to -2.7] — Crossvalidated; negative values mean that the fitted model performs worse than chance on the test set

7. Secondary Outcome: Antibody Titer Responses to Tetanus Booster Vaccine, Measured and Predicted Based on Early Post-vaccination Biomarkers in Healthy, Elderly Participants.
Description: Healthy elderly participants were simultaneously vaccinated at baseline with hepatitis vaccine, tetanus-diphtheria booster vaccine, and cholera vaccine. Antibody titers to tetanus were then measured 1 month after final vaccination, based on ELISA, and are defined as standardized "international units" of reactivity converted from optical densities, transformed to natural log (ln). In order to predict antibody responses blood samples were collected 7 days post-baseline vaccination to measure a wide variety of biomarkers by mRNA profiling, biochemical and flow cytometric assays. These biomarkers were then used in a machine-learning (random-forest based) model to predict antibody titers, transformed to natural log(ln).
Time Frame: Day 7 and 1 month after each final vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln International Units
Arm/Group | Elderly Participants
Number analyzed (Participants) | 143
ln International Units
  Predicted Titer | 1.43 (1.27)
  Measured Titer | 1.32 (1.84)
Statistical Analysis 1: Comparison: Elderly Participants; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Coefficient of Determination % = 23.7, 95% CI 2-sided [14.0 to 29.7] — Crossvalidated; negative values mean that the fitted model performs worse than chance on the test set

8. Secondary Outcome: Antibody Titer Responses to Reduced Diphtheria Toxin Vaccine, Measured and Predicted Based on Early Post-vaccination Biomarkers in Healthy, Elderly Participants.
Description: Healthy elderly participants were simultaneously vaccinated at baseline with hepatitis vaccine, tetanus-diphtheria booster vaccine, and cholera vaccine. Antibody titers to diphtheria were then measured 1 month after final vaccination, based on ELISA, and are defined as standardized "international units" of reactivity converted from optical densities, transformed to natural log (ln). In order to predict antibody responses blood samples were collected 7 days post-baseline vaccination to measure a wide variety of biomarkers by mRNA profiling, biochemical and flow cytometric assays. These biomarkers were then used in a machine-learning (random-forest based) model to predict antibody titers, transformed to natural log(ln).
Time Frame: Day 7 and 1 month after final vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln International Units
Arm/Group | Elderly Participants
Number analyzed (Participants) | 143
ln International Units
  Predicted Titer | -0.37 (1.36)
  Measured Titer | -0.46 (1.77)
Statistical Analysis 1: Comparison: Elderly Participants; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Coefficient of Determination % = 36.7, 95% CI 2-sided [28.7 to 41.5] — Crossvalidated;negative values mean that the fitted model performs worse than chance on the test set

9. Secondary Outcome: Antibody Titer Responses to Oral Cholera Vaccine (WC/rBS), Measured and Predicted Based on Early Post-vaccination Biomarkers in Healthy, Elderly Participants.
Description: Healthy elderly participants were simultaneously vaccinated at baseline with hepatitis vaccine, tetanus-diphtheria booster vaccine, and cholera vaccine. Antibody titers to cholera were then measured 3 weeks after final vaccination, based on ELISA, and are defined as standardized "international units" of reactivity converted from optical densities, transformed to natural log (ln). In order to predict antibody responses blood samples were collected 7 days post-baseline vaccination to measure a wide variety of biomarkers by mRNA profiling, biochemical and flow cytometric assays. These biomarkers were then used in a machine-learning (random-forest based) model to predict antibody titers, transformed to natural log(ln).
Time Frame: Day 7 and 3 weeks after final vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln International Units
Arm/Group | Elderly Participants
Number analyzed (Participants) | 143
ln International Units
  Predicted Titer | 5.24 (0.96)
  Measured Titer | 5.20 (1.55)
Statistical Analysis 1: Comparison: Elderly Participants; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Coefficient of Determination % = -2.2, 95% CI 2-sided [-7.8 to 4.4] — Crossvalidated; negative values mean that the fitted model performs worse than chance on the test set

ADVERSE EVENTS:
Groups:
- All Participants: Participants who received at least one dose of each vaccine
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/174
Other Adverse Events (participants affected / at risk) | 14/174
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=174)
Injection Site Pain (General disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.